CLINICAL TRIAL: NCT02907593
Title: Steroids and Surfactant in Extremely Low Gestation Age Infants Pilot Dose Escalation Trial
Brief Title: Steroids and Surfactant in Extremely Low Gestation Age Infants Dose Escalation Trial
Acronym: SASSIE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cynthia McEvoy (Other)
Collaborators: Thrasher Research Fund (Other); University of Florida (Other); Florida Hospital for Children (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Cynthia McEvoy, Principal Investigator, Professor of Pediatrics, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: SASSIE-001
Record Dates: First submitted 2016-08-02; First posted 2016-09-20 (Estimated); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Bronchopulmonary Dysplasia (BPD)
Keywords: Bronchopulmonary dysplasia; Pulmonary; Surfactant; Steroids; Extremely low gestational age
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Budesonide; calfactant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.025 mg/kg Budesonide (Experimental): 0.025 mg/kg Budesonide in Calfactant
  Interventions: Drug: Budesonide in Calfactant
- 0.050 mg/kg Budesonide (Experimental): 0.050 mg/kg Budesonide in Calfactant
  Interventions: Drug: Budesonide in Calfactant
- 0.10 mg/kg Budesonide (Experimental): 0.10 mg/kg Budesonide in Calfactant
  Interventions: Drug: Budesonide in Calfactant
- 0.15 mg/kg Budesonide (Experimental): 0.15 mg/kg Budesonide in Calfactant
  Interventions: Drug: Budesonide in Calfactant

INTERVENTIONS:
Drug: Budesonide in Calfactant — Budesonide in Calfactant
  Other Names: pulmicort respule; calfactant; budesonide; 0186-1986-04; infasurf

SUMMARY:
This is a phase I/II open-label study to determine the lowest, safe, effective dose of budesonide given with calfactant as the vehicle.

DETAILED DESCRIPTION:
This is a phase I/II open-label study to determine the lowest safe, effective dose of budesonide given with calfactant as the vehicle; the investigators will perform an unblinded dose escalation study. The investigators will administer four dosing levels of budesonide suspended in calfactant beginning with 0.025 mg/kg of budesonide administered to 8 extremely low gestational age newborns (ELGANs) who are intubated at 3-10 days of age. Daily doses (at the same dosage) will be administered to infants who remain intubated for a potential of 5 total doses in each patient. Subsequent groups of 8 infants each will receive 0.05 mg/kg, 0.10 mg/kg, and 0.15 mg/kg of budesonide in calfactant (up to 5 total doses in each patient). A total of up to 32 infants will be enrolled in the trial. The investigators will evaluate the clinical, laboratory and safety data from each group of treated infants to 28 days of age before moving to the next dosing level of budesonide.

ELIGIBILITY:
Inclusion Criteria:

1. > 23 0/7 and < 27 6/7 weeks of gestational age based on center's best estimate of due date (using earliest obstetrical ultrasound, last menstrual period, examination, and other pertinent available information)
2. Day of life 3-14 from the date and time of delivery, with the date of birth being DOL 0
3. Intubated and mechanically ventilated and do not anticipate extubation in next 24 hours

Exclusion Criteria:

1. Serious congenital malformations or chromosomal abnormality
2. Likely to be extubated in next 24 hours
3. Clinically unstable
4. Infants who have received systemic steroids prior to dosing with study medication.
5. Infants who have received Indocin, Ibuprofen, or acetaminophen ≤ 96 hours prior to enrollment window ending

Ages: 3 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia McEvoy, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Florida Hospital for Children, Orlando, Florida
  - Oregon Health ans Science University, Portland, Oregon
  - Vanderbilt Children's Hospital, Nashville, Tennessee

REFERENCES:
- [Background] Yeh TF, Chen CM, Wu SY, Husan Z, Li TC, Hsieh WS, Tsai CH, Lin HC. Intratracheal Administration of Budesonide/Surfactant to Prevent Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2016 Jan 1;193(1):86-95. doi: 10.1164/rccm.201505-0861OC. PMID 26351971
- [Background] Yeh TF, Lin HC, Chang CH, Wu TS, Su BH, Li TC, Pyati S, Tsai CH. Early intratracheal instillation of budesonide using surfactant as a vehicle to prevent chronic lung disease in preterm infants: a pilot study. Pediatrics. 2008 May;121(5):e1310-8. doi: 10.1542/peds.2007-1973. Epub 2008 Apr 21. PMID 18426851
- [Background] Roberts JK, Stockmann C, Dahl MJ, Albertine KH, Egan E, Lin Z, Reilly CA, Ballard PL, Ballard RA, Ward RM. Pharmacokinetics of Budesonide Administered with Surfactant in Premature Lambs: Implications for Neonatal Clinical Trials. Curr Clin Pharmacol. 2016;11(1):53-61. doi: 10.2174/1574884710666150929100210. PMID 26416605
- [Background] Barrette AM, Roberts JK, Chapin C, Egan EA, Segal MR, Oses-Prieto JA, Chand S, Burlingame AL, Ballard PL. Antiinflammatory Effects of Budesonide in Human Fetal Lung. Am J Respir Cell Mol Biol. 2016 Nov;55(5):623-632. doi: 10.1165/rcmb.2016-0068OC. PMID 27281349
- [Result] McEvoy CT, Ballard PL, Ward RM, Rower JE, Wadhawan R, Hudak ML, Weitkamp JH, Harris J, Asselin J, Chapin C, Ballard RA. Dose-escalation trial of budesonide in surfactant for prevention of bronchopulmonary dysplasia in extremely low gestational age high-risk newborns (SASSIE). Pediatr Res. 2020 Oct;88(4):629-636. doi: 10.1038/s41390-020-0792-y. Epub 2020 Feb 1. PMID 32006953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide | 0.15 mg/kg Budesonide
Started | 8 | 8 | 9 | 0 (Study ended prior to dosing level 4 (0.15 mg/kg).)
Completed | 8 | 8 | 8 | 0 (Study ended prior to dosing level 4 (0.15 mg/kg).)
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study ended prior to dosing level 4 (0.15 mg/kg).
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide | 0.15 mg/kg Budesonide | Total
Number analyzed (Participants) | 8 | 8 | 9 | 0 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 9 | 0 | 25
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: gestational age in weeks] | 25.3 (1.64) | 25.3 (1.25) | 24.4 (0.89) |  | 25.0 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 4 |  | 12
  Male | 6 | 2 | 5 |  | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 |  | 7
  Not Hispanic or Latino | 4 | 6 | 8 |  | 18
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 1 | 1 |  | 2
  White | 7 | 6 | 8 |  | 21
  More than one race | 0 | 1 | 0 |  | 1
  Unknown or Not Reported | 1 | 0 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 |  | 25
Number of participants that completed study [Count of Participants; unit: Participants] | 8 | 8 | 8 | 0 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of ELGANs With Clinical and Anti-inflammatory Efficacy of Escalating Doses of Budesonide Determined by Monitoring Respiratory Severity Score (RSS)
Description: Dose escalation will be defined as effective at the dose level in which 5 of 8 infants achieve the following:
  1. Extubation within 72 hours of first dose or after < 3 doses-without re-intubation before 28 days of age
  2. RSS on nasal continuous positive airway pressure (NCPAP) < 1.5 or on nasal cannula Fi02 <25% at < 2L/min at 28 days of age, persisting for at least 72 hours.
  3. Cumulative supplemental oxygen < 4.2 from time of enrollment to 28 days of age 4
  4. No respiratory support at 28 days, including no supplemental oxygen by nasal cannula
  AND a > 50% suppression of the tracheal aspirate interleukin-8 (IL-8) or CCL2 (chemokine ligand 2) at 24-72 hours (or prior to extubation if occurs at <24 hours after dosing) after the initial dose in 5 of 8 of the infants (this may be a different combination of 5 patients than those who met the above criteria).
Time Frame: 28 days of life for each dosing group
Population: Extremely low gestational age infants (ELGANs), born before 28 weeks gestation.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide | 0.15 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 8 | 0
Participants | 1 | 0 | 0 |

2. Primary Outcome: The Clinical and Anti-inflammatory Efficacy of Escalating Doses of Budesonide Suspended in Calfactant and Given Into the Lungs of ELGANs by Monitoring Tracheal Aspirate Cytokine Levels.
Description: Number of ELGANS with a clinical AND Cytokine response: a > 50% suppression of the tracheal aspirate interleukin-8 or chemokine ligand 2 at 24-72 hours (or prior to extubation if occurs at <24 hours after dosing) after the initial dose in 5 of 8 of the infants
Time Frame: 28 days of life for each dosing group
Population: No patient at the 0.025 mg/kg or at the 0.05 mg/kg or at the 0.10 mg/kg dosing level met the criteria for the primary outcome of a clinical and cytokine response. Due to this lack of response, we were approved by the Thrasher Foundation to not perform the dosing at the 0.15 mg/kg dosing level.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide | 0.15 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 8 | 0
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Adverse Events/Subject Safety
Description: Safety assessments will include the subject's vital signs, clinical laboratory testing, morbidities associated with prematurity, morbidities associated with administration of budesonide in calfactant, and Adverse Events (AE)s. Clinical parameters/ AEs of interest are those potentially consistent with elevated glucocorticoid levels and will be specifically evaluated. A Data and Safety Monitoring Board (DSMB) will be established to review safety data. All of the data will be reviewed to monitor subject safety.
Time Frame: Through 28 days of life
Population: No SAEs were considered to be treatment related.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 8
Participants | 8 | 8 | 8

4. Secondary Outcome: Serial Budesonide Levels, Peak
Description: The research team will obtain dried blood spot samples at 15 minutes, and 1 and 4 hours after the first dose of budesonide in calfactant for budesonide levels. Trough concentrations (Cmin) will be drawn before potential subsequent daily doses.
Time Frame: At 15 minutes, 1 and 4 hours after first dose and prior to each additional dose
Measure: Mean (54% Confidence Interval); unit: ng/mL
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 9
ng/mL | 7.70 [7.70 to 18.7] | 8.60 [7.70 to 18.7] | 18.7 [7.70 to 18.7]

5. Secondary Outcome: Serial Budesonide Levels, T 1/2
Description: as for outcome 4
Time Frame: At 15 minutes, 1 and 4 hours after first dose and prior to each additional dose
Measure: Mean (50% Confidence Interval); unit: h
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 9
h | 3.78 [3.20 to 3.78] | 3.20 [3.20 to 3.78] | 3.20 [3.20 to 3.78]

6. Secondary Outcome: Serial Budesonide Levels, AUC
Description: as for outcome 4
Time Frame: At 15 minutes, 1 and 4 hours after first dose and prior to each additional dose
Measure: Mean (48% Confidence Interval); unit: ng*h/mL
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 9
ng*h/mL | 39.4 [37.2 to 73.5] | 37.2 [37.2 to 73.5] | 73.5 [37.2 to 73.5]

7. Secondary Outcome: Respiratory Severity Score: Mean Airway Pressure and Oxygen Requirement at 28 Days of Age
Description: Clinical respiratory status (RSS and oxygen requirement) around dosing and at 28 days of age will be compared between dosing groups and also compared to the matched historical control patients from the "Trial of Late Surfactant:(TOLSURF) study.
  The respiratory severity score (RSS) is a simplified severity score consisting of the mean airway pressure (MAP) multiplied by the fraction of inspired oxygen (FiO2). This score ranges from 0 to 12, with a higher score indicating more severe disease.
Time Frame: 28 days of life for each dosing group
Measure: Mean (Standard Deviation); unit: Respiratory Severity Score
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide
Number analyzed (Participants) | 8 | 8 | 5
Respiratory Severity Score | 4.59 (3.74) | 4.94 (2.93) | 3.74 (2.97)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through 28 days of life.
Description: Adverse Event Definition:
  Any untoward medical occurrence in a patient or clinical investigation in which a subject is given a pharmaceutical product; does not necessarily have a causal relationship with such treatment, or Any unfavorable and unintended sign (including abnormal laboratory findings),symptom, or disease temporally associated with the use of a medicinal (investigational) product; not necessarily related to the product.
Arm/Group | 0.025 mg/kg Budesonide | 0.050 mg/kg Budesonide | 0.10 mg/kg Budesonide | 0.15 mg/kg Budesonide
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 3/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 4/9 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8 | 8/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.025 mg/kg Budesonide (N=8) | 0.050 mg/kg Budesonide (N=8) | 0.10 mg/kg Budesonide (N=9) | 0.15 mg/kg Budesonide (N=0)
Severe Respiratory Decompensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Necrotizing Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.025 mg/kg Budesonide (N=8) | 0.050 mg/kg Budesonide (N=8) | 0.10 mg/kg Budesonide (N=9) | 0.15 mg/kg Budesonide (N=0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated blood gas (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased urine output (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraventricular hemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Presumed formula aspiratiom (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reflux into ETT during dosing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PDA requiring treatment (Cardiac disorders) | 6 (6) | 5 (5) | 3 (3) | 0 (0)
Pulmonary decompensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Re-intubation during study (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Severe hypotension (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Severe respiratory decompensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Severe pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncontrolled hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of the study is not due to any safety concerns, but rather enrollment challenges and lack of response in patients. The FDA and IRB were notified and approved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02907593/Prot_SAP_000.pdf